CLINICAL TRIAL: NCT06199219
Title: Ex-Plissit Model Based Counseling on Sexual Function and Sexual Satisfaction in Women With Multiple Sclerosis: A Randomized Controlled Study
Brief Title: Ex-Plissit Model Based Counseling on Sexual Function and Sexual Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Vesile Koak, Dr., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21122023
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: MS (Multiple Sclerosis); Sexual Dysfunctions; Counseling
MeSH Terms: conditions — Multiple Sclerosis | interventions — Sex Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): Sexual counseling, based on the extended (EX-PLISSIT) model was offered to women for 6-10 weeks (until a solution was achieved).
  All interventions must begin with "Permission." Each stage of "Limited Information", "Special Recommendation" and "Intensive Therapy" is supported by "Allowing". Thus, the interaction between counselors and clients is improved
  Interventions: Other: Sexual counseling, based on the extended (EX-PLISSIT)
- Control Group (No Intervention): No intervention pretest posttest

INTERVENTIONS:
Other: Sexual counseling, based on the extended (EX-PLISSIT) — The EX-PLISSIT model is done in a cyclical manner. In other words, it is an interactive and repetitive model. All interventions must begin with "Permission." Each stage of "Limited Information", "Special Recommendation" and "Intensive Therapy" is supported by "Allowing". Thus, the interaction between counselors and clients is improved (Taylor and Davis 2006; Punjani and Papathanasoglu, 2019).
  Arms: Intervention Group

SUMMARY:
Aimed to determine the effect of sexual education based on the EX-PLISSIT model on sexual function and sexual satisfaction in women with multiple sclerosis.

The present study was a pretest-posttest randomized controlled study. Conducted between June and August 2023 in Turkey. The participants were MS patients who were women 18-49 years old. The intervention (n = 20) and a control group (n = 20). The intervention group received sexual counseling based on the EX-PLISSIT model. The model consists of four levels. The levels are permission, limited information, specific suggestions and intensive therapy. Counseling was presented in six to eight sessions according to the women's sexual problems. The Female Sexual Function Index (FSFI) and the New Sexual Satisfaction Scale were used to measure the sexual function and sexual satisfaction of the participants.

Data were analyzed using the Statistical Package for the Social Sciences (SPSS) version 21. P values below 0.05 were considered statistically significant.

DETAILED DESCRIPTION:
Within the scope of this research, sexual counseling, based on the extended (EX-PLISSIT) model was offered to women for 6-10 weeks (until a solution was achieved). The EX-PLISSIT model is based on the core concepts of the PLISSIT model. The PLISSIT model is an effective, convenient and cost effective counseling method. This model was designed by Annon (1976) and includes the stages permission, limited ınformation, specific recommendations and intensive therapy. It is known that the PLISSIT model is effective for SD. The PLISSIT Model has been updated and expanded because it offers one-way, passive interaction. While counseling is linear in the PLISSIT model, it is feedback-oriented in the EX-PLISSIT model. This is one of the reasons why the EX-PLISSIT model is superior to the PLISSIT model. Unlike PLISSIT's linear mode; The EX-PLISSIT model is done in a cyclical manner. In other words, it is an interactive and repetitive model. All interventions must begin with "Permission." Each stage of "Limited Information", "Special Recommendation" and "Intensive Therapy" is supported by "Allowing". Thus, the interaction between counselors and clients is improved. While in the PLISSIT model, a direct transition can be made from one step to another, in the EX-PLISSIT model, the permission stage is at the center of the other stages and techniques such as review, and examination are used to increase the client's self-awareness. The EX-PLISSIT model is a practical guide for nursing research and practice.

ELIGIBILITY:
Inclusion Criteria:

Being between the reproductive age range of 18-49

* Being sexually active for at least 1 year
* MS diagnosis must have been confirmed at least 6 months ago
* EDSS scale score <7
* Be willing to participate
* Not having any chronic disease (thyroid problems, diabetes mellitus, cardiovascular diseases, etc.)
* Being able to speak and understand Turkish

Exclusion Criteria:

* Pregnant or breastfeeding women
* Those who score 16 and above according to the BECK depression scale
* Women under treatment for sexual dysfunction
* Women with inadequate cognitive levels
* Having an MS attack within the last month
* Alcohol and drug addiction

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The Female Sexual Function Index (FSFI) Score | 8 weeks
  The Female Sexual Function Index 19-item self-report questionnaire evaluating the sexual functions of female patients. The questions are regarding women's sexual feelings and responses during the last four weeks. Accordingly, the highest score that can be obtained from the scale is 36.0 and the lowest score is 2.0.

SECONDARY OUTCOMES:
New Sexual Satisfaction Scale (NSSS) Score | 8 weeks
  The New Sexual Satisfaction Scale (NSSS) was developed by Štulhofer et al. (2010), and the psychometric properties of the Turkish form were examined by Tuğut (2016). Turkish NSSS is a valid and reliable measurement tool to evaluate sexual satisfaction in Turkish women.

CONTACTS AND LOCATIONS:
Overall Officials: Vesile Kocak, Study Chair — Necmettin Erbakan University
Locations (1):
- Vesile KOÇAK, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided